CLINICAL TRIAL: NCT06191770
Title: Comparison of Morphine With Nalbuphine in a Multimodal Approach for Pain Relief in Patients Undergoing Gynecological Procedures: Randomized Controlled Double Blinded Clinical Trial
Brief Title: Comparison of Morphine With Nalbuphine in a Multimodal Approach for Pain Relief in Patients Undergoing Gynecological Procedures: Randomized Controlled Double Blind Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, BAL CHAND, BAL CHAND, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-0209-414
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Morphine; Nalbuphine

STUDY DESIGN:
Intervention Model Description: Two groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind Clinical Trial, CTU prepare the Medications, and Patient, investigator and Data Collector was completely blind to the Stuidy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morphine Arm (Active Comparator): NRS score used
  Interventions: Procedure: Morphine,
- Nalbuphine Arm (Active Comparator): Both Groups
  Interventions: Procedure: Morphine,

INTERVENTIONS:
Procedure: Morphine, — Nalbuphine along multimodal analgesia(Paracetamol and Ketamine)
  Other Names: Nalbuphine

SUMMARY:
This study was conducted in the Aga Khan University Hospital, Karachi. Pakistan is developing country and overall shortage of Morphine in developing country.

Rationalizing, in multimodal analgesia, Nalbuphine is equivalent to morphine in open Abdominal hysterectomy

DETAILED DESCRIPTION:
A large number of patients undergoing major surgical procedures need gold standard analgesic like morphine for adequate pain control. Shortage of Morphine results in inadequate pain relief leading to delayed recovery, prolonged hospitalization and persistent post-surgical pain syndrome.

For better surgical outcome, there is a strong need to find an alternative to morphine in a multi modal analgesia that help optimize pain relief with less opioids in patients undergoing gynecological procedures

ELIGIBILITY:
Inclusion Criteria:

* All ASA I and ASA II women, age b/w 18-59 scheduled for Elective open moderate to major gynecological procedures at Aga Khan University Hospital

Exclusion Criteria:

* Patient is unwilling to participate or provide informed consent History of chronic pain or pain syndrome with concurrent opioid medication use Fibromyalgia Patient has received opioids and/or tramadol in the past 4 hours History of adverse reaction to morphine, ketamine and nalbuphine Presence of oxygen dependent pulmonary disease, liver cirrhosis or renal disease requiring dialysis.

Presence of Ischemic heart disease Presence of intracranial mass or vascular lesion. Presence of psychosis or hallucinations Weight greater than 115kg or less than 45 kg

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only Females
Enrollment: 66 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Morphine Versus Nalbuphine in a multimodal Analgesia for Patients undergoing Gynecological Procedures: A double blind randomized controlled trial | 1 year
  The primary objective was to compare the analgesic requirement of morphine with nalbuphine in multimodal approach (with Paracetamol and Ketamine).

SECONDARY OUTCOMES:
Morphine Versus Nalbuphine in a multimodal Analgesia for Patients undergoing Gynecological Procedures: A double blind randomized controlled trial | 1 year
  To assess the adverse events associated with nalbuphine and morphine.

CONTACTS AND LOCATIONS:
Locations (1):
- Gauhar Afshan, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
we can shaire study protocol, if anyone required
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: Anyone